CLINICAL TRIAL: NCT01046643
Title: Hormones and Cognitive Processing in Early Postmenopausal Women
Brief Title: Early Menopause Hormone Treatment and Cognition
Acronym: R21
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Yolanda Smith, M.D., Professor, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R21AG031951-01A1 (NIH); 1R21AG031951-01A1 (NIH)
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Results first posted 2014-05-19 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Menopausal Syndrome
Keywords: Women; Healthy; Menopausal; Hormone treatment
MeSH Terms: interventions — Estradiol; Progesterone; Annexin A2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Estrogen followed by Placebo (Active Comparator): Estrogen treatment with Estradiol (E2) followed by Placebo.
  Interventions: Drug: Estradiol (E2); Drug: Progesterone (P10) x10
- Progesterone followed by Placebo (Active Comparator): Progesterone (P10) treatment followed by Placebo.
  Interventions: Drug: Progesterone (P10) x90
- Placebo followed by Estrogen (Active Comparator): Placebo followed by Estrogen treatment with Estradiol (E2)
  Interventions: Drug: Estradiol (E2); Drug: Progesterone (P10) x10
- Placebo followed by Progesterone (Active Comparator): Placebo followed by Progesterone (P10) treatment.
  Interventions: Drug: Progesterone (P10) x90

INTERVENTIONS:
Drug: Estradiol (E2) — One Estradiol capsule (1mg) once a day, at the same time each day, for 90 days; followed by one Progesterone (200mg) once a day, at the same time each day, for 10 days to slough endometrial lining; followed by one Placebo capsule once a day, at the same time each day, for 90 days.
  Other Names: E2
  Arms: Estrogen followed by Placebo; Placebo followed by Estrogen
Drug: Progesterone (P10) x90 — One Progesterone capsule (200mg) once a day, at the same time each day, for 90 days; followed by one Placebo capsule (to mirror Progesterone capsule to slough endometrial lining in Estradiol recipients) once a day, at the same time each day, for 10 days ; followed by one Placebo capsule once a day, at the same time each day, for 90 days.
  Other Names: P10
  Arms: Placebo followed by Progesterone; Progesterone followed by Placebo
Drug: Progesterone (P10) x10 — One Progesterone (200mg) capsule once a day for 10 days, to slough endometrial lining for patients taking Estradiol. Patients taking Progesterone will take an equivalent Placebo capsule during this time period.
  Other Names: P10
  Arms: Estrogen followed by Placebo; Placebo followed by Estrogen

SUMMARY:
The objective of this study is to evaluate the neurobiological effects of hormone therapy (HT) in healthy early postmenopausal women. The studies proposed in this project seek to define the association between different hormone forms (estradiol only and progesterone only) versus placebo on brain functional measures. The functional measures will include the performance of the volunteers on a comprehensive neuropsychological testing battery, and the brain functional responses to episodic memory (verbal and non-verbal) challenges as well as emotional processing determined with functional magnetic resonance imaging (fMRI).

DETAILED DESCRIPTION:
Specific Aims

Aim 1. To examine the effects of estradiol alone on brain functioning in early post-menopausal women during verbal and non-verbal cognitive tasks.

Hypothesis: It is expected that with estradiol treatment brain activation will be more prominent in the hippocampus and prefrontal cortical areas compared to placebo. The magnitude of activation in these regions will be positively correlated with task performance in the scanner and with the results of neuropsychological tests assessing verbal and non-verbal delayed recall.

Aim 2. To determine the effects of progesterone alone on brain functioning in early postmenopausal women during verbal and non-verbal cognitive tasks.

Hypothesis: It is expected that with progesterone treatment brain activation in the hippocampus and prefrontal cortical areas will be decreased compared to both the placebo condition (within subjects) and the estradiol condition (between subjects). Interindividual variations in the magnitude of activation in these regions will be positively correlated with task performance in the scanner and with the results of neuropsychological tests assessing verbal and non-verbal delayed recall.

Aim 3. To determine the individual effects of estradiol and progesterone on brain functioning in early postmenopausal women during emotional processing stimuli.

Hypothesis: During negative stimuli estradiol-treated women compared to placebo group, are expected to have increased activity in the amygdala, posterior cingulate, and orbitofrontal cortex, while in progesterone-treated women compared to placebo, decreased activity is expected in these brain regions.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* Ages 45-55, 6 - 36 months from their last menstrual period.

Exclusion Criteria:

* Left handedness
* Acute medical illness
* Neurologic illness
* Psychiatric illness
* Heart disease
* Thromboembolic disease
* Liver disease
* Uncorrected thyroid disease
* Diabetes
* Neurological disease
* Porphyria
* Allergy to estradiol
* Progesterone or lactose
* Lactose intolerance
* Claustrophobia
* Contraindications to MRI (including pacemakers, surgical clips or metallic surgical devices)
* Smoking within the last 3 years
* Use of hormones within the last 3 months
* Current or past history of substance abuse
* History of head injury or loss of consciousness
* Medications with actions on the central nervous system
* Endometrial lining greater than 5mm
* Ovarian pathology on ultrasound
* Abnormal mammogram
* Migraines
* Fasting cholesterol >300 mg/dl, and fasting triglycerides >300 mg/dl
* Creatinine level > 1.5 mg/dl
* Aspartate transaminase (AST) or Alanine transaminase (ALT) greater than two times the top normal range
* Follicle stimulating hormone (FSH) values <40 IU/L
* estradiol >40 pg/ml.
* Subjects with HAM-D score > 8, HAM-A > 6 during screening will not be eligible.

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yolanda R. Smith, M.D., Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: +++__Women were recruited from 3/1/2010 to 7/29/2011 through local newspaper ads, flyers, electronic newsletters, bulletin boards, clinics and the Women's Health Registry, a University of Michigan database of women interested in participating in women's health related clinical research.
Pre-assignment Details: Several enrolled participants were excluded from the trial prior to assignment in groups on the basis of the risk factors identified at the pre-screening appointment. Some others did not qualify due to their lab results which did not meet the inclusion criteria.
Groups:
- Estrogen Followed by Placebo: Estrogen treatment with Estradiol (E2)
  One Estradiol capsule (1mg) once a day, at the same time each day, for 90 days followed by one Placebo capsule once per day for 90 days, at the same time each day
- Progesterone Followed by Placebo: Progesterone (P10) treatment
  One Progesterone (P10) (200 mg) capsule once a day, at the same time each day, for 90 days, followed by one Placebo capsule once per day for 90 days, at the same time each day.
- Placebo Followed by Estrogen: One Placebo capsule once per day for 90 days, at the same time each day, followed by one Estradiol capsule (E2) (1mg) once a day, at the same time each day, for 90 days.
- Placebo Followed by Progesterone: One Placebo capsule once per day for 90 days, at the same time each day, followed by one Progesterone (P10) (200 mg) capsule once a day, at the same time each day, for 90 days.
Period: First Period Treatment or Placebo
Arm/Group | Estrogen Followed by Placebo | Progesterone Followed by Placebo | Placebo Followed by Estrogen | Placebo Followed by Progesterone
Started | 9 | 7 | 7 | 7
Completed | 9 | 6 | 7 | 7
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Period: Washout Period
Arm/Group | Estrogen Followed by Placebo | Progesterone Followed by Placebo | Placebo Followed by Estrogen | Placebo Followed by Progesterone
Started | 9 | 6 | 7 | 7
Completed | 9 | 6 | 7 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Second Period Treatment or Placebo
Arm/Group | Estrogen Followed by Placebo | Progesterone Followed by Placebo | Placebo Followed by Estrogen | Placebo Followed by Progesterone
Started | 9 | 6 | 7 | 7
Completed | 9 | 6 | 7 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Estrogen and Placebo: Estrogen treatment with Estradiol (E2)
  Participants received both an Estradiol capsule (E2) (1mg) and a Placebo capsule in a randomized sequence (for a total of two sequences of 90 days each, consisting of one capsule, once per day at the same time each day).
- Progesterone and Placebo: Progesterone treatment (P10)
  Participants received both a Progesterone capsule (P10) (200 mg) and a Placebo capsule in a randomized sequence (for a total of two sequences of 90 days each, consisting of one capsule, once per day at the same time each day).
- Total: Total of all reporting groups
Arm/Group | Estrogen and Placebo | Progesterone and Placebo | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (2.2) | 51.2 (2.9) | 51.5 (2.5)
Gender [Number; unit: participants]
  Female | 9 | 7 | 16
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 7 | 16
Months since Last Menstrual Period [Mean (Standard Deviation); unit: months] | 19.81 (9.57) | 16.69 (9.80) | 18.41 (9.63)
Education [Mean (Standard Deviation); unit: years] | 15.75 (2.82) | 17.19 (2.67) | 16.4 (2.8)
Estradiol [Mean (Standard Deviation); unit: pg/mL] | 17.75 (6.30) | 14.38 (6.25) | 16.24 (6.40)
Follicle-Stimulating Hormone [Mean (Standard Deviation); unit: mIU/mL] | 92.34 (33.85) | 80.86 (21.60) | 87.19 (29.11)
BMI [Mean (Standard Deviation); unit: kg/m²] | 27.13 (6.13) | 28.38 (3.8) | 27.69 (5.17)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Brain Activation Patterns in Verbal Tasks Determined With the Functional Magnetic Resonance Imaging (fMRI) Scans
Description: Measure the changes in brain activity in verbal tasks with hormone use (either estradiol or progesterone) versus placebo.
  The test is a deep and shallow verbal processing task, where the subjects are presented lists of words, one word at a time, and are asked to make one of 2 decisions about each list. One decision is whether each word is written in upper or lower case letters (shallow processing), and the other decision is whether each word denotes an abstract or concrete concept (deep processing).
  The test was administered 3 months after baseline and 38 weeks after baseline.
Time Frame: August 2010 - March 2012
Population: Within the Estrogen/Placebo groups, 3 participants were unable to complete the needed fMRI analyses due to adverse events, and in the Progesterone/Placebo groups, 1 participant's fMRI scans were damaged and unable to be used in the analysis.
Measure: Mean (Standard Deviation); unit: percent BOLD signal changes
Groups:
- Estrogen: Estrogen treatment with Estradiol (E2)
  Estradiol (E2) : One Estradiol capsule (1mg) once a day, at the same time each day, for 90 days
- Progesterone: Progesterone treatment
  Progesterone (P10) : One Progesterone (200 mg) capsule once a day, at the same time each day, for 90 days
- Placebo (Estrogen): Placebo phase of Estradiol (E2) treatment
  One Placebo capsule once a day, at the same time each day, for 90 days
- Placebo (Progesterone): Placebo phase of Progesterone (P10) treatment
  One Placebo capsule once a day, at the same time each day, for 90 days
Arm/Group | Estrogen | Progesterone | Placebo (Estrogen) | Placebo (Progesterone)
Number analyzed (Participants) | 13 | 12 | 13 | 12
percent BOLD signal changes
  Medial Frontal Cortex | .14 (.12) | .13 (.16) | .05 (021) | .13 (.18)
  Left Hippocampus | -.04 (.14) | -.01 (.15) | -.13 (.16) | .09 (.34)
  Right Hippocampus | -.06 (.18) | -.06 (.13) | -.14 (.16) | .01 (.24)
Statistical Analysis 1: Comparison: Estrogen vs Placebo (Estrogen); Category = Medial Frontal Cortex p-value for null hypothesis = <0.05; Test type: Superiority or Other; p = .222, t-test, 2 sided — Category = Medial Frontal Cortex
Statistical Analysis 2: Comparison: Estrogen vs Placebo (Estrogen); Category = Left Hippocampus p-value for null hypothesis = <0.05; Test type: Superiority or Other; p = .107, t-test, 2 sided — Category = Left Hippocampus
Statistical Analysis 3: Comparison: Estrogen vs Placebo (Estrogen); Category = Right Hippocampus p-value for null hypothesis = <0.05; Test type: Superiority or Other; p = .127, t-test, 2 sided — Category = Medial Frontal Cortex
Statistical Analysis 4: Comparison: Progesterone vs Placebo (Progesterone); Category = Medial Frontal Cortex p-value for null hypothesis = <0.05; Test type: Superiority or Other; p = .954, t-test, 2 sided — Category = Medial Frontal Cortex
Statistical Analysis 5: Comparison: Progesterone vs Placebo (Progesterone); Category = Left Hippocampus p-value for null hypothesis = <0.05; Test type: Superiority or Other; p = .385, t-test, 2 sided — Category = Left Hippocampus
Statistical Analysis 6: Comparison: Progesterone vs Placebo (Progesterone); Category = Right Hippocampus p-value for null hypothesis = <0.05; Test type: Superiority or Other; p = .310, t-test, 2 sided — Category = Right Hippocampus

2. Secondary Outcome: Neuropsychological Testing Scores - Verbal Learning Retention
Description: Changes in neuropsychological testing measures (verbal learning retention) with hormone use (either estradiol or progesterone) versus placebo.
  Subjects are given tests that present them with a series of words. They are asked to recall how many items they can remember, and then some time later, are asked to recall the items again. The retention measure is how many items they can remember at the later time point, compared to the earlier time point. Adapted from the Benton Visual Memory Test, Revised.
  The tests were administered 3 months after baseline and 38 weeks after baseline.
Time Frame: August 2010 - March 2012
Population: Within the Estrogen/Placebo groups, 3 participants were unable to complete the needed fMRI analyses due to adverse events, and in the Progesterone/Placebo groups, 1 participant's fMRI scans were damaged.
Measure: Mean (Standard Deviation); unit: percent retention
Arm/Group | Estrogen | Progesterone | Placebo (Estrogen) | Placebo (Progesterone)
Number analyzed (Participants) | 13 | 12 | 13 | 12
percent retention | 96.79 (6.72) | 97.12 (15.30) | 94.94 (10.75) | 98.44 (12.25)
Statistical Analysis 1: Comparison: Estrogen vs Placebo (Estrogen); p-value for null hypothesis = <0.05; Test type: Superiority or Other; p = .594, t-test, 2 sided
Statistical Analysis 2: Comparison: Progesterone vs Placebo (Progesterone); p-value for null hypothesis = <0.05; Test type: Superiority or Other; p = .653, t-test, 2 sided

3. Primary Outcome: Changes in Brain Activation Patterns in Visual Tasks Determined With the Functional Magnetic Resonance Imaging (fMRI) Scans
Description: Measure the changes in brain activity in visual tasks with hormone use (either estradiol or progesterone) versus placebo.
  The test is a visual working memory task, where the women are presented with 3 geometric grids on the screen. The target grid is on top, and 2 test grids are on the bottom. The women must decide if the right or left test grid matches the grid on top. There are 3 conditions: a match condition where all 3 grids are shown simultaneously, and 2 delay conditions, where the target grid is shown first, disappears, and the test grids appear after a 1 or a 4 second delay.
  The test was administered 3 months after baseline and 38 weeks after baseline.
Time Frame: August 2010 - March 2012
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent BOLD signal changes
Arm/Group | Estrogen | Progesterone | Placebo (Estrogen) | Placebo (Progesterone)
Number analyzed (Participants) | 13 | 12 | 13 | 12
percent BOLD signal changes
  Medial Frontal Cortex | .25 (.17) | .47 (.28) | .16 (.41) | .20 (.43)
  Left Hippocampus | .21 (.20) | .38 (.25) | .23 (.38) | .21 (.29)
  Right Hippocampus | .29 (.17) | .38 (.29) | .21 (.48) | .15 (.29)
Statistical Analysis 1: Comparison: Estrogen vs Placebo (Estrogen); Category = Medial Frontal Cortex p-value for null hypothesis = <0.05; Test type: Superiority or Other; p = .452, t-test, 2 sided — Category = Medial Frontal Cortex
Statistical Analysis 2: Comparison: Estrogen vs Placebo (Estrogen); Category = Left Hippocampus p-value for null hypothesis = <0.05; Test type: Superiority or Other; p = .868, t-test, 2 sided — Category = Left Hippocampus
Statistical Analysis 3: Comparison: Progesterone vs Placebo (Progesterone); Category = Right Hippocampus p-value for null hypothesis = <0.05; Test type: Superiority or Other; p = .549, t-test, 2 sided — Category = Right Hippocampus
Statistical Analysis 4: Comparison: Progesterone vs Placebo (Progesterone); Category = Medial Frontal Cortex p-value for null hypothesis = <0.05; Test type: Superiority or Other; p = .124, t-test, 2 sided — Category = Medial Frontal Cortex
Statistical Analysis 5: Comparison: Progesterone vs Placebo (Progesterone); Category = Left Hippocampus p-value for null hypothesis = <0.05; Test type: Superiority or Other; p = .158, t-test, 2 sided — Category = Left Hippocampus
Statistical Analysis 6: Comparison: Progesterone vs Placebo (Progesterone); Category = Right Hippocampus p-value for null hypothesis = <0.05; Test type: Superiority or Other; p = .055, t-test, 2 sided — Category = Right Hippocampus

4. Secondary Outcome: Neuropsychological Testing Scores - Visual Learning Retention
Description: Changes in neuropsychological testing measures (visual learning retention) with hormone use (either estradiol or progesterone) versus placebo.
  Subjects are given tests that present them with a series of pictures. They are asked to recall how many items they can remember, and then some time later, are asked to recall the items again. The retention measure is how many items they can remember at the later time point, compared to the earlier time point. Adapted from the California Verbal Learning Test - 2nd edition.
  The tests were administered 3 months after baseline and 38 weeks after baseline.
Time Frame: August 2010 - March 2012
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent retention
Arm/Group | Estrogen | Progesterone | Placebo (Estrogen) | Placebo (Progesterone)
Number analyzed (Participants) | 13 | 12 | 13 | 12
percent retention | 93.31 (19.22) | 97.59 (13.67) | 97.01 (14.79) | 96.19 (12.06)
Statistical Analysis 1: Comparison: Estrogen vs Placebo (Estrogen); p-value for null hypothesis = <0.05; Test type: Superiority or Other; p = .561, t-test, 2 sided
Statistical Analysis 2: Comparison: Progesterone vs Placebo (Progesterone); p-value for null hypothesis = <0.05; Test type: Superiority or Other; p = .726, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Estrogen Followed by Placebo: Estrogen treatment with Estradiol (E2)
  One Estradiol capsule (E2) (1mg) once a day, at the same time each day, for 90 days followed by one Placebo capsule once per day for 90 days, at the same time each day.
- Progesterone Followed by Placebo: Progesterone treatment
  One Progesterone (P10) (200 mg) capsule once a day, at the same time each day, for 90 days, followed by one Placebo capsule once per day for 90 days, at the same time each day.
- Placebo Followed by Estrogen: One Placebo capsule once per day for 90 days, at the same time each day, followed by one Estradiol capsule (E2) (1mg) capsule once a day, at the same time each day, for 90 days.
Arm/Group | Estrogen Followed by Placebo | Progesterone Followed by Placebo | Placebo Followed by Estrogen | Placebo Followed by Progesterone
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/7 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 1/9 | 1/7 | 3/7 | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Estrogen Followed by Placebo (N=9) | Progesterone Followed by Placebo (N=7) | Placebo Followed by Estrogen (N=7) | Placebo Followed by Progesterone (N=7)
Claustrophobia (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Side effects of hormone use (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No